CLINICAL TRIAL: NCT06983067
Title: A Prospective, Open-label, Single-Arm Study Evaluating the Sentire C1000 Surgical Robotic System in Ureteral Reconstruction for Benign Ureteral Strictures
Brief Title: Application of the Sentire C1000 for Ureteral Stricture Repair
Acronym: ROBUST-C1000
Status: Recruiting | Type: Observational
Sponsor: Xuesong Li (Other)
Responsible Party: Sponsor-Investigator, Xuesong Li, Peking University First Hospital, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: F-00882-001
Record Dates: First submitted 2025-05-04; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Ureteral Stricture; Hydronephrosis
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Simple anastomosis reconstruction group: Including pyeloplasty, stenectomy and reanastomosis, and bladder reimplantation
  Interventions: Device: Cornerstone C1000 Robotic Surgery System
- Patch Repair Group: Includes oral mucosa, appendix patches, etc.
  Interventions: Device: Cornerstone C1000 Robotic Surgery System
- Intestinal/ileal Substitute Ureteral Group: These include the ileal substitution ureter and colonic substitution ureter procedures.
  Interventions: Device: Cornerstone C1000 Robotic Surgery System

INTERVENTIONS:
Device: Cornerstone C1000 Robotic Surgery System — Minimally invasive surgical instruments are controlled by the physician using a master-slave operating system for urologic laparoscopic surgical operations.

SUMMARY:
The purpose of this clinical study is to evaluate the safety and efficacy of the Sten® Laparoendoscopic Surgical System C1000 for benign ureteral reconstruction surgery. This is a single-arm, open-label, prospective, non-randomized cohort study.

Eligibility criteria for recruitment to this study included how to include labeling: (1) patients aged ≥18 years and ≤80 years, male and female; (2) patients who need to undergo upper urinary tract repair surgery; (3) patients who are suitable for ureteral reconstruction surgery as confirmed by the investigator; (4) subjects voluntarily participating in the clinical trial and agreeing to, or their guardian agreeing to, and signing an informed consent form; (5) willingness to cooperate with and complete the trial follow-up and related examinations. The research subjects of this project were recruited openly, and the patients were enrolled after being informed of the study-related information, risks and benefits by the project participants and then screened to meet the enrollment criteria. A total of 50 patients will be enrolled.

The study objectives and endpoints include the following: primary endpoints: (1) the rate of surgical non-referral (2) the success rate of surgical treatment; secondary endpoints: (1) the loading time (2) the operating time of the surgeon (3) the estimated intraoperative blood loss (4) the postoperative patient's pain scores (5) the evaluation of the physiological load of the surgeon (6) the evaluation of the mental load of the surgeon (7) the rate of intraoperative transfusion (8) the duration of the hospital stay after the operation (9) the evaluation of physician satisfaction (9) the evaluation of physician's satisfaction). (9) Physician satisfaction rating (10) Overall postoperative complication rate (11) Adverse events and serious adverse events (12) Device defects (13) Postoperative readmission rate (14) Reoperation rate (15) Mortality rate.

The expected overall duration is 9 months, with an expected enrollment time of 6 months and a subject follow-up time of approximately 3 months.

DETAILED DESCRIPTION:
The purpose of this clinical study is to evaluate the safety and efficacy of the Sten® Laparoendoscopic Surgical System C1000 for benign ureteral reconstruction surgery. This is a single-arm, open-label, prospective, non-randomized cohort study.

Eligibility criteria for recruitment to this study included how to include labeling: (1) patients aged ≥18 years and ≤80 years, male and female; (2) patients who need to undergo upper urinary tract repair surgery; (3) patients who are suitable for ureteral reconstruction surgery as confirmed by the investigator; (4) subjects voluntarily participating in the clinical trial and agreeing to, or their guardian agreeing to, and signing an informed consent form; (5) willingness to cooperate with and complete the trial follow-up and related examinations. The research subjects of this project were recruited openly, and the patients were enrolled after being informed of the study-related information, risks and benefits by the project participants and then screened to meet the enrollment criteria. A total of 50 patients will be enrolled.

The study objectives and endpoints include the following: primary endpoints: (1) the rate of surgical non-referral (2) the success rate of surgical treatment; secondary endpoints: (1) the loading time (2) the operating time of the surgeon (3) the estimated intraoperative blood loss (4) the postoperative patient's pain scores (5) the evaluation of the physiological load of the surgeon (6) the evaluation of the mental load of the surgeon (7) the rate of intraoperative transfusion (8) the duration of the hospital stay after the operation (9) the evaluation of physician satisfaction (9) the evaluation of physician's satisfaction). (9) Physician satisfaction rating (10) Overall postoperative complication rate (11) Adverse events and serious adverse events (12) Device defects (13) Postoperative readmission rate (14) Reoperation rate (15) Mortality rate.

The expected overall duration is 9 months, with an expected enrollment time of 6 months and a subject follow-up time of approximately 3 months.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients aged ≥18 years and ≤80 years, male or female; (2) Patients who need to undergo upper urinary tract repair surgery; (3) Patients who are suitable for ureteral reconstruction as confirmed by the investigator; (4) Subjects who voluntarily participate in the clinical trial and agree or whose guardians agree and sign the informed consent form; (5) Willing to cooperate and complete the trial follow-up and related examinations.

Exclusion Criteria:

* (1) Presence of severe drug/imaging contrast allergy; (2) Patients with a history of pelvic/abdominal surgery and assessed for extensive severe adhesions; (3) Those with a previous history of other malignancies and judged by the investigator to be unsuitable for enrollment; (4) Diseases that are not expected to tolerate pneumoperitoneum or prolonged head-down-foot-up position, or diseases that do not allow intraoperative positioning, such as spinal deformity or ankylosing spondylitis; (5) Those with serious comorbidities (heart, lung, liver, brain, kidney and other diseases) and those who are physically weak and cannot tolerate general anesthesia or surgery; (6) Those with serious bleeding tendency or coagulation disorders; (7) Patients who have been using anticoagulant or antiplatelet aggregating drugs for a long time, or those who have stopped using anticoagulant or antiplatelet aggregating drugs for less than 1 week before surgery (except for the prophylactic use of low molecular heparin before surgery); (8) Patients with active infectious diseases or other severe non-infectious infections; (9) Those who are positive for Human Immunodeficiency Virus (HIV), Hepatitis B Surface Antigen (Hepatitis B) or Hepatitis C Surface Antigen (Hepatitis C).

Hepatitis B Surface Antigen (HbsAg)-positive, Hepatitis C Virus (HCV)-positive, and syphilis-positive patients; (10) Persons with severe allergies, suspected or confirmed alcohol, drug or drug addiction; (11) Those with a history of epilepsy or psychosis or with cognitive impairment; (12) Women who are pregnant, breastfeeding, or planning to become pregnant during the trial, or male or female patients who do not wish to use barrier contraception during the trial; (13) Participation in any other clinical trial (except non-interventional trials) within 3 months prior to signing the informed consent form, planning to undergo any other major surgical procedure during the trial, or inability to recover from the side effects of a previous procedure; (14) Any other circumstances that the investigator considers inappropriate for participation in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility criteria for enrollment in this study included how to include labeling: (1) patients aged ≥18 years and ≤80 years, male and female; (2) patients who need to undergo upper urinary tract repair surgery; (3) patients who are suitable for ureteral reconstruction as confirmed by the investigator; (4) subjects voluntarily participating in the clinical trial and agreeing to, or whose guardian agrees to, and signing an informed consent form; (5) willingness to cooperate with and complete the trial follow-up and related examinations.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Surgical non-transfer rate | During the surgery
  Surgical non-transfer rate is defined as failure to switch from the test medical device (Laparoendoscopic Surgical System) assisted approach to other surgical device control system assisted, laparoscopic surgery or open surgery.
  Surgical non-referral rate = number of subjects whose surgery was not referred/total number of subjects x 100%.
Success rate of surgical treatment | 3 months postoperatively
  At 3 months postoperatively, surgical treatment was considered successful when the following conditions were also met:
  * No ureteral obstruction on investigator-assessed imaging and no deterioration/progression of renal function from baseline.
  * No interventions (endoluminal dilatation, surgical interventions, etc.) for disease progression or recurrence after study treatment, except for interventions for complications of the surgery Success rate of surgical treatment = number of subjects with successful surgical treatment/total number of subjects × 100%.

SECONDARY OUTCOMES:
Installation time | During the surgery
  Defined as starting with the push of the patient-side robot and pushing to the bedside until all arms are aligned with the cannula and the arms are adjusted to the proper position. Unit: minutes.
Surgeon operating time | During the surgery
  Defined as the time from the first effective movement of the arm by the surgeon until the surgeon completes the surgical procedure and the arm stops moving (excluding pause time due to force majeure). Unit: minutes.
  The starting point of the operation time: the first effective movement of the operating arm controlled by the surgeon; the end point: the surgeon completes the surgical operation and the movement of the operating arm stops.
Estimated blood loss | During the surgery
  Defined as intraoperative blood loss, i.e., the estimated total blood loss from the time the test medical device enters the body cavity incision to the completion of the surgical incision suture, including the blood volume in the suction bottle and intraoperative gauze, etc., and excluding intraoperative irrigation fluid or perfusion fluid, etc., with 1g counted as 1mL. unit: mL.
Postoperative patient pain scores | During the surgery
  At the screening/baseline period, at the 24±4h postoperative follow-up, and at the 3-month postoperative follow-up, subjects were assessed for postoperative pain according to a visual analogue scale (VAS) ranging from a score of 0 (no pain) to a score of 10 (maximum pain).
Evaluation of intraoperative physiologic load by the surgeon | During the surgery
  On the day of surgery, the Localized Discomfort Experience Scale was taken to evaluate the surface electromyography of the muscles of the shoulder, neck, upper extremity, and lumbar region.
  Calculation formula: the primary surgeon's intraoperative physiologic load score = the sum of the primary surgeon's intraoperative physiologic load score for all subjects ÷ the number of cases of subjects undergoing surgical treatment.
Wise Load Evaluation of the Surgeon | During the surgery
  On the day of surgery, the Subjective Mental Load Scale was taken for evaluation.
  Calculation formula: subjective surgeon's surgical mental load score = sum of all subjects' subjective surgeon's surgical mental load scores ÷ number of cases of subjects undergoing surgical treatment.
Intraoperative blood transfusion rates | During the surgery
  Defined as the number of subject cases requiring blood transfusion as a percentage of the total number of subject cases from the first surgical incision to the completion of suturing of the last surgical incision.
Post-operative hospitalization time | Perioperative period
  Defined as the total number of days the subject was hospitalized from the day of surgery to discharge, which was recorded at follow-up.
Physician satisfaction ratings | During the surgery
  The investigators rated the performance and comfort level of the test medical devices through a questionnaire after completing the procedure.

OTHER OUTCOMES:
Overall complication rate at 3 months postoperatively | 3 months postoperatively
  Complications were recorded from the first intraoperative incision to the 3-month postoperative follow-up, and the overall complication rate was evaluated by the Clavien-Dindo grading system (Clavien-Dindo grading of 1 or higher).
Adverse events | 3 months postoperatively
  To evaluate the type, incidence (%), and frequency (number of events) of adverse events and device-related adverse events during the study period.
Serious adverse event | 3 months postoperatively
  To evaluate the type, incidence (%), and frequency (number of events) of serious adverse events and device-related serious adverse events during the study period.
Instrument defects | During the surgery
  To evaluate the type, incidence (%), and frequency (number of events) of device defects during the study period.
Post-operative readmission rate | 3 months postoperatively
  To evaluate the incidence (%) and frequency of readmission from the time the subject was discharged to 3 months postoperatively.
Reoperation rate | 3 months postoperatively
  The incidence (%) and frequency of reoperation within 3 months after surgery were evaluated.
Mortality rate | 3 months postoperatively
  To evaluate the incidence (%) and frequency of subject deaths within 3 months postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No